CLINICAL TRIAL: NCT02684045
Title: A Retrospective Review of Charts to Assess Outcomes in Subjects That Received MAGNIFUSE® DBM in the Posterolateral Lumbar Spine
Brief Title: Retrospective Chart Review to Assess Outcomes in Subjects That Received MAGNIFUSE® in the Posterolateral Lumbar Spine
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-03
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Subjects Received MAGNIFUSE in Posterolateral Lumbar Spine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this chart review is to assess outcomes in subjects that received MAGNIFUSE in the posterolateral lumbar spine at 1 or 2 continuous levels from L1-S1.

ELIGIBILITY:
Inclusion Criteria:

A subject's medical record must contain the following for the subject to be included:

1. Posterolateral surgical procedure using MAGNlFUSE with local autograft and/or iliac crest bone graft at one or two continuous lumbar levels from L1-S1.
2. Radiographs available for fusion assessment by clinician at 12 and/or 24 month post-surgery visits.
3. Subject must be at least 18 years old at the time of index procedure.

Exclusion Criteria:

The subject data will be excluded from this study if the medical record indicates:

1. Additional surgical treatment adjacent to the initial lumbar levels treated per Inclusion Criterion 1.
2. Infection at index level(s) at time of surgery.
3. Extant tumor (evident at any level), spinal metastasis, or spinal tumor at the time of surgery.
4. Pregnant at time of surgery.
5. Surgery is due to trauma (e.g., motor vehicle accident or high impact fall).
6. Use of growth factors or growth peptide (BMP2, BMP7, or iFactor) in the index-level fusion surgery.
7. Procedure is a revision surgery for previously failed fusion at the surgery index level(s).
8. Subjects with body mass index > 40 at the time of surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who underwent a posterolateral surgical procedure with MAGNIFUSE in the lumbar spine.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Fusion status at 12 or 24 months | 12 or 24 months
  Fusion status will be assessed using the Lenke posterior fusion criteria below:
  * Grade I: Solid trabeculated transverse process and facet fusions bilaterally.
  * Grade II: Thick fusion mass on one side, and difficult to visualize on the other side.
  * Grade III: Suspected lucency or defect in the fusion mass.
  * Grade IV: Definite resorption of graft with fatigue of instrumentation.

SECONDARY OUTCOMES:
Back pain and leg pain measured by visual analog scale (VAS) | 12 or 24 months
Pain and Disability status measured by Oswestry Disability Index (ODI) | 12 or 24 months
Quality of life measured by EQ-5D | 12 or 24 months

OTHER OUTCOMES:
complications of interest | 12 or 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Midwest Ortho. Center, Peoria, Illinois
  - University of Virginia, Charlottesville, Virginia